CLINICAL TRIAL: NCT04068129
Title: Performance of Two Photoscreeners With Enhanced Housing
Brief Title: Enhanced Housing Photoscreeners 2WIN and GoCheckKids Compared in Burma and Alaska
Status: Completed | Type: Observational
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: ABCD GCK Kaleidos
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-08

CONDITIONS: Amblyopia; Anisometropia
MeSH Terms: conditions — Amblyopia; Anisometropia | interventions — Refraction, Ocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Burma: Patients from remote Burma clinic
  Interventions: Device: photoscreen
- Alaska: Patients in pediatric ophthalmology clinic
  Interventions: Device: photoscreen

INTERVENTIONS:
Device: photoscreen — Determine amblyopia risk factors
  Other Names: refraction

SUMMARY:
"Adaptica" (Padova, Italy) designed a fixed-distance, dark portable tube with power and remote control for the "2WIN: photoscreener. GoChecksKids designed a flash-concentrating case for the iPhone 7+ to more quickly achieve two-axis photoscreen. These devices were compared to confirmatory exams in children and young adults in a remote Burma clinic and in an Alaskan pediatric ophthalmology practice.

DETAILED DESCRIPTION:
Photoscreening with follow up confirmatory exams for referred and passed interpretations were offered to children and young adults at a remote clinic in the Karen State of eastern Burma (Myanmar). The clinic had intermittent 220 Volt power generator, but no internet or cell phone coverage.

Consecutive patients in a "WiFi-equipped" pediatric ophthalmology practice in Anchorage, Alaska had photoscreening before confirmatory examination.

Each patient had photoscreening with the "2WIN" photoscreener installed in the "Kaleidos" housing. In Anchorage, the devise was controled by the wireless tablet computer. In Burma, however, despite a "WiFi router" not connected to internet, the tablet computer would not connect to the 2WIN and therefore the "Kaleidos" read-trap door was opened so the 2WIN could be activated and controlled manually. The" 2WIN" stored results on an "micro-SD" memory card which was eventually downloaded to computer.

Each patient also had photoscreening with GoCheckKids (GCK) on an "iPhone 7 Plus" using the enhanced, flash-concentrating cell-phone case. In Anchorage, in addition to on-site smart-phone interpretation, images were uploaded to the central reading center for secondary interpretation. In Burma, all images were retained on the smart phone and eventually uploaded for GoCheckKids central secondary analysis after return to urban internet availability. In Burma, a portable, light-wieght tent was used to provide a dim screening environment with less distraction.

Confirmatory exams were performed consistent with 2003 and 2013 American Association for Pediatric Ophthalmology and Strabismus (AAPOS) uniform guidelines. Cycloplegic refractions were performed 20-40 minutes after cyclopentolate 1% instillation. Visual acuity was checked with patched, surround "HOTV" at 3 meters threshold with at least 3 of 4 optotypes correct. Validation was performed with conventional 2 x 2 screen-exam matrix, and also with Alaska Blind Child Discovery (ABCD) 3 x 3 matrix including inconclusive results (no instrument interpretation or unable to gain a reading) with inconclusive interpretations considered a referral.

ELIGIBILITY:
Inclusion Criteria:

* at least one eye

Exclusion Criteria:

* bilateral enucleation

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and young adults attending eye clinics in Burma and Alaska
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Amblyopia Rick Factor prevalence | February 15, 2019 through April 16, 2019
  AAPOS 2003 and 2013 defined ARFs

SECONDARY OUTCOMES:
Refractive Error | February 15, 2019 through April 16, 2019
  Glasses prescription

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Arnold, MD, Principal Investigator — Alaska Blind Child Discovery
Locations (1):
- Alaska Children's EYE & Strabismus, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data on ABCD website
Supporting Information: CSR
Time Frame: Fall 2019
Access Criteria: ongoing
URL: http://www.abcd-vision.org/references/index.html

REFERENCES:
- [Background] Martin SJ, Htoo HE, Hser N, Arnold RW. Performance of Two Photoscreeners Enhanced by Protective Cases. Clin Ophthalmol. 2020 May 25;14:1427-1435. doi: 10.2147/OPTH.S251451. eCollection 2020. PMID 32546951
- Available data/document: Individual Participant Data Set — http://www.abcd-vision.org/references/index.html